CLINICAL TRIAL: NCT00226720
Title: Comparison of Efficacy of an Outpatient vs Inpatient Detoxification Program for Alcohol Dependent Patients Seeking Abstinence. A Prospective Randomized Clinical Trial.
Brief Title: Outpatient Versus Inpatient Detoxification Program for Alcohol Dependent Patients Seeking Abstinence: The IN/OUT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Direction Générale de la Santé, France (Other)
Responsible Party: Myriem TOUHAMI-CARRIER, Department Clinical Research of the Developpement
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: P000807; AOM98176
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2007-04

CONDITIONS: Alcoholism; Alcohol Dependence
Keywords: alcoholism; Alcohol dependence; Detoxification; Abstinence maintain; Efficacy; Ambulatory detoxification
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): at the hospital
  Interventions: Procedure: Outpatient detoxification program
- 2 (Active Comparator): out of the hospital
  Interventions: Procedure: Outpatient detoxification program

INTERVENTIONS:
Procedure: Outpatient detoxification program — Outpatient detoxification program

SUMMARY:
Detoxification, in an inpatient or outpatient program, is the primary and essential step for managing alcohol dependence. The superiority of one or other method of detoxification has never been proved in several previous randomized clinical trials (RCT). The aim of this multicenter RCT was to compare efficiency, on the abstinence rate as the primary outcome, at 1 and 3 months follow-up of two alcohol detoxification programs (a 5/7-days inpatient detox vs. an ambulatory detox).

DETAILED DESCRIPTION:
Among patients consulting in 4 alcohol treatment centers in France seeking treatment for withdrawal, we included those who met criteria for current alcohol-dependence (DSM IV) and having drinking during the past three days before randomization. Exclusion criteria were: patients' refusal of one or other method, contraindication for outpatient detoxification method (history of DELIRIUM TREMENS or withdrawal seizures), homelessness, Major Depressive Episode assessed by MADRS > 25, current Substance Abuse Disorder (except nicotine), indication for hospitalization (severe somatic disorder), judicial injunction, family crisis, patients seeking antabuse treatment.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol dependence according to DSM IV
* Detoxification program requested by patients

Exclusion Criteria:

* Refusal of the patient for the hospitalization or ambulant weaning alcoholic
* contraindication in ambulant weaning
* The state of the patient requires a hospitalization
* Ask of the patient for a treatment by the ESPERAL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2002-09; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Abstinence rate at 3 Months & 6 Months follow-up. Abstinence is defined as no alcohol drinking during the period between the last day of the detoxification program and the evaluation. | at 3 Months & 6 Months

SECONDARY OUTCOMES:
Relapse rate. Relapse is defined as drinking more than 4 Units per occasion (3 for women) and more than one occasion per week during the 6 months follow-up after the last day of detoxification program. | during the 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Philippe M. BATEL, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- BEAUJON Hospital, Clichy, France

REFERENCES:
- [Background] Limosin F, Romo L, Batel P, Ades J, Boni C, Gorwood P. Association between dopamine receptor D3 gene BalI polymorphism and cognitive impulsiveness in alcohol-dependent men. Eur Psychiatry. 2005 May;20(3):304-6. doi: 10.1016/j.eurpsy.2005.02.004. PMID 15935433
- [Background] Batel P, Reynaud-Maurupt C, Lavignasse P, Constant MV, Kopp P, Jourdain JJ, Videau B, Mucchielli A, Riff B, Lowenstein W. [Risk factors of early drop-out during induction of high-dose buprenorphine substitution therapy. A study of 1085 opiate addicts]. Presse Med. 2004 Oct 23;33(18 Suppl):5-9. doi: 10.1016/s0755-4982(04)72375-1. French. PMID 15617169
- [Background] Batel P, Balester-Mouret S. [Care network in addictive pathologies: where is it?]. Rev Prat. 2003 Jun 15;53(12):1335-9. French. PMID 12920943
- [Background] Pessione F, Ramond MJ, Peters L, Pham BN, Batel P, Rueff B, Valla DC. Five-year survival predictive factors in patients with excessive alcohol intake and cirrhosis. Effect of alcoholic hepatitis, smoking and abstinence. Liver Int. 2003 Feb;23(1):45-53. doi: 10.1034/j.1600-0676.2003.01804.x. PMID 12640727
- [Background] Gorwood P, Limosin F, Batel P, Hamon M, Ades J, Boni C. The A9 allele of the dopamine transporter gene is associated with delirium tremens and alcohol-withdrawal seizure. Biol Psychiatry. 2003 Jan 1;53(1):85-92. doi: 10.1016/s0006-3223(02)01440-3. PMID 12513948
- [Background] Lavignasse P, Lowenstein W, Batel P, Constant MV, Jourdain JJ, Kopp P, Reynaud-Maurupt C, Riff B, Videau B, Mucchielli A. Economic and social effects of high-dose buprenorphine substitution therapy. Six-month results. Ann Med Interne (Paris). 2002 May;153(3 Suppl):1S20-6. PMID 12218879
- [Background] Batel P, Michaud P. [Risky alcohol drinking or problems and brief interventions]. Gastroenterol Clin Biol. 2002 May;26(5 Suppl):B158-62. No abstract available. French. PMID 12068283
- [Background] Gorwood P, Aissi F, Batel P, Ades J, Cohen-Salmon C, Hamon M, Boni C, Lanfumey L. Reappraisal of the serotonin 5-HT(1B) receptor gene in alcoholism: of mice and men. Brain Res Bull. 2002 Jan 1;57(1):103-7. doi: 10.1016/s0361-9230(01)00641-4. PMID 11827742
- [Background] Gorwood P, Limosin F, Batel P, Duaux E, Gouya L, Ades J. The genetics of addiction: alcohol-dependence and D3 dopamine receptor gene. Pathol Biol (Paris). 2001 Nov;49(9):710-7. doi: 10.1016/s0369-8114(01)00236-x. PMID 11762133
- [Background] Batel P, Lariviere P. [Late-onset alcohol withdrawal syndrome]. Ann Med Interne (Paris). 2000 Oct;151 Suppl B:B27-9. French. PMID 11104941
- [Background] Gorwood P, Batel P, Ades J, Hamon M, Boni C. Serotonin transporter gene polymorphisms, alcoholism, and suicidal behavior. Biol Psychiatry. 2000 Aug 15;48(4):259-64. doi: 10.1016/s0006-3223(00)00840-4. PMID 10960156
- [Background] Batel P. Addiction and schizophrenia. Eur Psychiatry. 2000 Mar;15(2):115-22. doi: 10.1016/s0924-9338(00)00203-0. PMID 10881208
- [Background] Gorwood P, Batel P, Gouya L, Courtois F, Feingold J, Ades J. Reappraisal of the association between the DRD2 gene, alcoholism and addiction. Eur Psychiatry. 2000 Mar;15(2):90-6. doi: 10.1016/s0924-9338(00)00207-8. PMID 10881204
- [Background] Batel P. [Alcohol withdrawal syndrome in the hospital]. Rev Prat. 1999 Feb 15;49(4):387-90. French. PMID 10319688
- [Background] Quinones-Jenab V, Batel P, Schlussman SD, Ho A, Kreek MJ. Cocaine impairs maternal nest building in pregnant rats. Pharmacol Biochem Behav. 1997 Dec;58(4):1009-13. doi: 10.1016/s0091-3057(97)00311-0. PMID 9408207
- [Background] Batel-Copel LM, Kornblith AB, Batel PC, Holland JC. Do oncologists have an increasing interest in the quality of life of their patients? A literature review of the last 15 years. Eur J Cancer. 1997 Jan;33(1):29-32. doi: 10.1016/s0959-8049(96)00414-5. PMID 9071895
- [Background] Batel P. A critique of chapter 3: "Individual drinking and degree of risk". Addiction. 1995 Nov;90(11):1450-1. doi: 10.1111/j.1360-0443.1995.tb02804.x. No abstract available. PMID 8528027
- [Background] Batel P. The treatment of alcoholism in France. Drug Alcohol Depend. 1995 Sep;39 Suppl 1:S15-21. doi: 10.1016/0376-8716(95)01169-y. PMID 8565793
- [Background] Batel P, Pessione F, Maitre C, Rueff B. Relationship between alcohol and tobacco dependencies among alcoholics who smoke. Addiction. 1995 Jul;90(7):977-80. doi: 10.1046/j.1360-0443.1995.90797711.x. PMID 7663320
- [Background] Batel P, Pessione F, Bouvier AM, Rueff B. Prompting alcoholics to be referred to an alcohol clinic: the effectiveness of a simple letter. Addiction. 1995 Jun;90(6):811-4. doi: 10.1046/j.1360-0443.1995.9068118.x. PMID 7633298